CLINICAL TRIAL: NCT03347097
Title: The Safety and Efficacy Study of Autologous Tumor-infiltrating T Lymphocyte（TIL）and Transgenic Modified TIL Cells Adoptive Therapies for Patients With Glioblastoma Multiforme
Brief Title: Adoptive Cell Therapy of Autologous TIL and PD1-TIL Cells for Patients With Glioblastoma Multiforme
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Huashan Hospital (Other)
Collaborators: Shanghai Cell Therapy Research Institute (Other)
Responsible Party: Principal Investigator, Yu Yao, MD, Resident, Huashan Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2017-241
Record Dates: First submitted 2017-11-02; First posted 2017-11-20 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Glioblastoma Multiforme
Keywords: glioma; TIL; PD1-TIL; immunotherapy
MeSH Terms: conditions — Glioblastoma; Glioma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TIL cells (Experimental): 10 days after the end of chemotherapy or radiotherapy，the 300ml TIL cells ( TIL saline + 0.25% human serum albumin) was injected intravenously 2 times every 30 days .
  Interventions: Drug: TIL
- PD1-TIL cells (Experimental): 10 days after the end of chemotherapy or radiotherapy，the 300ml PD1-TIL cells ( PD1-TIL saline + 0.25% human serum albumin) was injected intravenously 2 times every 30 days .
  Interventions: Drug: PD1-TIL

INTERVENTIONS:
Drug: TIL
  Arms: TIL cells
Drug: PD1-TIL
  Arms: PD1-TIL cells

SUMMARY:
At present, the investigators want to evaluate safety and efficacy of cell therapy based on Tumor-infiltrating T Lymphocyte (TIL）in glioblastoma. Here, we also constructed a transgenic modified TIL cells, stablely express a high-level full-length PD1 antibody (PD1-TIL cells), which can transduce signals to activate T cells and result in tumor killing. In this study, we design two group patients treated with TIL cells and PD1-TIL cells respectively to determine the safety and efficacy of autologous TILs or genetically modified TILs in patients with glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

1. Recurrent patients with histologically confirmed brain glioblastoma multiforme.
2. Patients with maximum safe resection of the tumor (≥95%) confirmed with contrast MR or CT within 72 hours after surgery.
3. Age from 18 to 70 years.
4. Karnofsky performance score ≥ 60.
5. Adequate organ function within 14 days of study registration including the following: Adequate bone marrow reserve: absolute neutrophil (segmented and bands) count, (ANC) ≥ 1.0×10^9/L, platelets ≥100×10^9/L; hemoglobin ≥ 9 g/dL. Hepatic: bilirubin ≤1.3 mg/dL or 0-22 mmol/L, aspartate transaminase (AST) and alanine transaminase (ALT) < 3×upper limit of normal (ULN). Renal: Normal serum Creatinine for age (below) or creatinine clearance >60 ml/min/1.73 m2. Electrocardiogram: normal.
6. Written informed consent must be obtained from all patients.

Exclusion Criteria:

1. Pregnant or breast-feeding patients. Pregnancy testing will be performed on all menstruating females within 14 days of study enrollment.

   Patients with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements.
2. Patients with history of immune system abnormalities such as hyperimmunity (e.g., autoimmune diseases) and hypoimmunity (e.g., myelodysplastic disorders, marrow failures, AIDS, ongoing pregnancy, transplant immuno-suppression), or medication of cortisol.
3. Patients with any conditions that could potentially alter immune function (e.g., AIDS, multiple sclerosis, diabetes, renal failure).

Patients currently received any other investigational agents.

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events related to TIL and PD1-TIL cells infusion | 1 month

SECONDARY OUTCOMES:
Treatment Responses Rate | 6 months
Overall Survival Rate | 24 months
Progression-free Survival Rate | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No